# Evaluation of the Effects of Silk and Polyester Suture on Postoperative Complications in Lower Impacted Third Molar Teeth Surgery

Levent Ciğerim DDS, PhD <sup>1</sup>, Mehmet Güzel<sup>1</sup>, Abdulrahman Alghalaeini<sup>1</sup>, Zeynep Dilan Orhan <sup>1</sup> Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Van, TURKEY

# Corresponding author: Levent Ciğerim

Address: Van Yüzüncü Yıl University, Faculty of Dentistry, Department of Oral and Maxillofacial

Surgery, Van, Turkey Postal Code: 65080

E-mail address: levent139@hotmail.com Phone:+905321633287 Office Phone: 904322251744

Fax: +904322251747

#### Levent CİĞERİM

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery levent139@hotmailmail.com, +905321633287, <a href="https://orcid.org/0000-0001-5218-8568">https://orcid.org/0000-0001-5218-8568</a>

#### Mehmet GÜZEL

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery dtmehmetguzel@gmail.com, +905363609854, https://orcid.org/0000-0002-9621-0496

#### Abdulrahman Alghalaeini

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery dentist.a.gh@gmail.com, +905355524762, https://orcid.org/0000-0002-0443-5592

### Zeynep Dilan Orhan

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery <a href="mailto:reynequal-tom">reynequal-tom</a>, +905425525525, <a href="https://orcid.org/0000-0003-1333-9073">https://orcid.org/0000-0003-1333-9073</a>

# **Study Protocol, Methods and Procedures**

The study is planned to be performed on 30 patients who will apply to Van Yüzüncü Yıl University, Faculty of Dentistry, Department of Oral, Dental and Maxillofacial Surgery, who will have impacted lower wisdom teeth extracted.

Silk suture (4/0 Neosilk Ultra Silk 19mm 3/8 hoop) will be used on one side of the patients, and polyester suture (4-0 Ticron Blue 18" P-12 Cutting, Coviden Sutur) will be used on the other side. 3/8 diameter, reverse sharp in groups. 4/0 thick sutures with needles will be used. When the patients first apply to the clinic, their anamnesis will be taken and their panoramic images will be taken after their clinical evaluations. It will be determined whether the individuals have lower impacted wisdom teeth or not.

Individuals aged 18 and over, individuals without systemic disease, bilaterally similar positions will be used. Individuals with impacted lower wisdom teeth and individuals with an operation time of 30 minutes or less will be included. Pregnant and lactating individuals, individuals who do not come to their postoperative controls, individuals who use different drugs than those recommended, and individuals who are allergic to the study drugs and the suture materials to be used will be excluded from the study.

In this randomized, single-blind, split-mouth study, evaluations will be made for all patients with preoperative face measurements (for evaluation of swelling) and maximum mouth opening (for evaluation of trismus). The mentioned measurements and evaluations will be repeated on the 2nd and 7th postoperative days. In addition, postoperative pain will be evaluated with the VAS scale, which will be filled in by the patients themselves. The same surgical procedure will be performed by the same surgeon for all patients. After local anesthesia (2ml, 80 mg Articaine hydrochloride + 0.02mg Epinephrine bitartrate), a 3-corner flap containing the vertical incision passing through the mesial of the number 7 will be lifted, the bone will be removed under saline cooling, and the teeth will be separated when necessary. Afterwards, the extraction sockets will be irrigated with saline, bleeding will be controlled and the area will be closed primarily with silk or polyester suture material. All patients will receive postoperative analgesics (1200mg Ibuprofen daily tablet 2\*1) and antiseptic mouthwash (0.15% Benzydamine hydrochloride and 0.12% Chlorhexidine gluconate 3\*1). The obtained data will be evaluated statistically.

## **Statistical Data Analysis**

Deviation, Minimum and Maximum values; will be expressed as numbers and percentages for categorical variables. Mann-Whitney U analysis will be used to compare group means in terms of continuous independent variables. In addition, the Wicoxon test will be calculated in the comparison of double dependent groups. In order to determine the relationship between these variables, Spearman correlation coefficients will be calculated separately for the groups. Chi-square test will be used to determine the relationship between groups and categorical variables. Statistical significance level will be taken as 5% in calculations and SPSS statistical package program will be used for calculations.